CLINICAL TRIAL: NCT03374124
Title: The Surgical Prognosis Based Diagnostic Strategy for Eosinophilic Chronic Rhinosinusitis: A Retrospective Study
Brief Title: The Surgical Prognosis Based Diagnostic Strategy for Eosinophilic Chronic Rhinosinusitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jianbo Shi (Other)
Responsible Party: Sponsor-Investigator, Jianbo Shi, Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: 20171019
Record Dates: First submitted 2017-11-27; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Sinusitis; Nasal Polyps
Keywords: Chronic rhinosinusitis; Eosinophil; Surgery; Diagnosis
MeSH Terms: conditions — Sinusitis; Nasal Polyps; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The samples were abtained during endoscopic sinus surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- postoperational CRS: observe the symptoms and endoscopic appearance
  Interventions: Diagnostic Test: sinonasal outcome test-22

INTERVENTIONS:
Diagnostic Test: sinonasal outcome test-22 — Evaluate the nasal mucosal inflammation condition and overall quality-of-life of CRS patients
  Other Names: Lund-Kennedy endoscopic score

SUMMARY:
Previous studies have demonstrated that the eosinophilic inflammation of nasal mucosa is associated with the uncontrolled condition of chronic rhinosinusitis after surgery. However, the definition of the eosinophilic chronic rhinosinusitis is not very clear. Japanese researchers have designed a scoring system to diagnose eosinophilic chronic rhinosinusitis. In this study, the investigators hope to examine the practicability of this scoring system and have a better knowledge of eosinophilic chronic rhinosinusitis in china.The retrospective study was conducted in a tertiary hospital. Participants received functional endoscopic sinus surgery more than 1 years were called back for evaluation. A diagnosis cut off value of eosinophil count was determined by the surgery prognosis. Then different factors were compared between participants with eosinophilic CRS and those with non-eosinophilic CRS to establish the appropriated diagnosis approach for eosinophilic CRS.

DETAILED DESCRIPTION:
The retrospective study was conducted in a tertiary hospital. Participants received functional endoscopic sinus surgery more than 1 years were called back for evaluation. A diagnosis cut off value of eosinophil count was determined by the surgery prognosis. Then different factors were compared between participants with eosinophilic CRS and those with non-eosinophilic CRS to establish the appropriated diagnosis approach for eosinophilic CRS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis according to European position paper of rhinosinusitis and nasal polyps 2007.

Exclusion Criteria:

* Immunodeficiency diseases, history of head and/or facial trauma, cancer or organ transplant recipients.
* Pregnancy or lactation.
* Acute respiratory tract infection within one month before the study.
* Patients without pathological samples.
* Antrochoanal polyp and cyst of the paranasal sinuses.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic rhinosinusitis patients after endoscopic surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
nasal symptoms | through study completion, an average of 2 year
  presence of bothersome congestion or rhinorrhea or olfactory loss or headache.(VAS more than 7 points).
endoscopic appearance indicate the uncontrol of CRS | through study completion, an average of 2 year
  The presence of diseased mucosa (nasal polyps, mucopurulent secretions,and/or inflamed mucosa) under endoscopy.
  (Lund-kennedy endoscopic score: Polyp≥1 or Oedema≥2 or Discharge≥2; 0-Absence of polyps;1-polyps in middle meatus only;2-polyps beyond middle meatus but not blocking the nose completely;3-polyps completely obstructing the nose.
  Oedema: 0-absent; 1-mild; 2-severe.Discharge: 0-no discharge; 1-clear, thin discharge; 2-thick, purulent discharge.)

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Shi, doctor, Study Director — Ent department, the first affiliated hospital, Sun Yat-sen University
Locations (1):
- the first affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong, China